CLINICAL TRIAL: NCT02991456
Title: Phase II Randomized Study to Evaluate Efficacy, Patient Satisfaction, and Compliance of the Oral Combination of Rolapitant (Varubi®) Plus Ondansetron vs. Ondansetron Monotherapy in Malignant Glioma Patients Receiving Radiotherapy (RT) and Concomitant Temozolomide
Brief Title: Rolapitant as an Antiemetic in Malignant Glioma Patients Receiving Radiotherapy and Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00076418
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Chemo-radiation Induced Nausea and Vomiting
Keywords: malignant glioma; temozolomide; temodar; radiation; emesis; nausea; vomiting; chemotherapy; Affronti; Peters; 00076418
MeSH Terms: conditions — Vomiting; Glioma; Nausea | interventions — rolapitant; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A (Active Comparator): Daily ondansetron alone for 3 weeks, followed by the use of rolapitant (one dose on day 22) plus continued daily ondansetron for 3 weeks.
  Interventions: Drug: Rolapitant; Drug: Ondansetron
- Sequence B (Active Comparator): Single dose of rolapitant (one dose on day 1) plus daily ondansetron for 3 weeks, followed by daily ondansetron alone for 3 weeks.
  Interventions: Drug: Rolapitant; Drug: Ondansetron

INTERVENTIONS:
Drug: Rolapitant — single 180 mg dose by mouth
  Other Names: Varubi
Drug: Ondansetron — 8 mg by mouth daily
  Other Names: Zofran

SUMMARY:
The purpose of this phase 2 study is to assess the efficacy and patient satisfaction of oral rolapitant plus ondansetron vs. oral ondansetron monotherapy in malignant glioma (MG) patients receiving standard of care radiation (RT) and temozolomide (TMZ) therapy. This is a randomized phase 2 trial of rolapitant plus ondansetron vs. ondansetron monotherapy for the prevention of chemo-radiation induced nausea and vomiting in primary MG subjects receiving RT and concomitant multi-dose TMZ.

DETAILED DESCRIPTION:
All eligible subjects should receive a planned total dose of 54-60 gray (GY) of radiation and 75 mg/m2 of TMZ daily for a total of six weeks. Patients will be randomized to receive one of two antiemetic treatment sequences: sequence A that involves administration of ondansetron alone for 3 weeks followed by a single dose of rolapitant (day 22) plus daily ondansetron for 3 weeks or sequence B that involves a single dose of rolapitant (day 1) plus daily ondansetron for 3 weeks followed by 3 weeks of daily ondansetron alone. The study has one primary endpoint: complete response (CR) rate. Participation in this study may result in reduced chemo-radiation induced nausea and vomiting, however, risks include the common side effects of rolapitant including decreased appetite, neutropenia, dizziness, dyspepsia, urinary tract infection, stomatitis, and anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed, newly-diagnosed malignant glioma (glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligoastrocytoma, anaplastic pleomorphic xanthoastrocytoma, or anaplastic oligodendroglioma) and are scheduled to receive radiotherapy (for a total of 54-60 Gy) and concomitant daily temozolomide therapy (at a dose of 75 mg/m^2 for one complete 6-week cycle).
* Age ≥ 18 years
* Karnofsky ≥ 60% or ECOG 0-2
* Hematocrit >29%, Absolute Neutrophil Count >1,000 cells/mm^3, platelets >100,000 cells/mm^3
* Serum creatinine <1.4 mg/dl, bilirubin <1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN. For subjects with known liver metastases ≤ 5 x ULN, and alanine aminotransferase (ALT) ≤ 2.5 x ULN. For subjects with known liver metastases ≤ 5 x ULN
* For patients on higher than physiological level of corticosteroids, they must have been on a stable dose for 1 week prior to initiating study drug, and the dose should not be escalated over entry dose level, if clinically possible
* Ability and willingness to give informed consent
* Female patients of childbearing potential must have a negative pregnancy test at Screening
* Female patients of childbearing potential must agree to use an acceptable method of birth control from the signing of informed consent and to continue its use during the study and for at least 90 days after the final dose
* Male patients must agree to use an acceptable form of birth control from study Day 1 through at least 90 days after the final dose

Exclusion Criteria:

* Co-medications that may interact with rolapitant as reviewed by Duke Preston Robert Tisch Brain Tumor investigator pharmacist.
* Co-medications that are contraindicated in patients on rolapitant including pimozide, thioridazine, carbamazepine, colchicine, dabigatran (Pradaxa), edoxaban (Savaysa), fosphenytoin, metoprolol, phenobarbital, phenytoin, primidone, and warfarin
* Inability or unwillingness to cooperate with the study procedures
* Prophylactic medication for the prevention of nausea and vomiting 24 hours prior to the start of radiation therapy through the full course of radiation therapy is prohibited, with the exception of the study drug. Corticosteroids will be allowed for treatment of cerebral swelling
* Previous participation in any clinical trial involving rolapitant
* Any vomiting, retching, dry heaves, or clinically significant nausea (i.e., NCI Common Toxicity Criteria version 4.0 grade 2-4 nausea) caused by any etiology in the 24 hrs. preceding day 1 of the study intervention (ondansetron or ondansetron with rolapitant) as scheduled to begin on day 1 of radiation and chemotherapy. Or a patient who has a history of anticipatory nausea and vomiting.
* Ongoing vomiting from any organic etiology
* Received rolapitant within 21 days prior to study enrollment
* Prior cancer chemotherapy or radiotherapy
* Any current treatment, medical history, or uncontrolled condition, other than malignancy, (e.g., alcoholism or signs of alcohol abuse, seizure disorder, medical or psychiatric condition) that, in the opinion of the investigator, would confound the results of the study or pose any unwarranted risk in administering study drug to the subject
* Patient has a known hypersensitivity to the administration of rolapitant or its excipients
* Patient has a history of severe renal or hepatic impairment, severe bone marrow suppression, or systemic infection
* Patient is a woman with a positive serum pregnancy test at Screening, is pregnant, breast-feeding, or is planning to conceive children within the projected duration of the study treatment
* Patient has taken the following agents within the last 48 hours prior to the start of treatment with study drug:
* 5-HT3 antagonists (ondansetron, granisetron, dolasetron, tropisetron, etc.).
* Benzamides (metoclopramide, alizapride, etc.)
* Domperidone
* Cannabinoids
* Natural Killer (NK)-1 antagonist (aprepitant)
* Benzodiazepines (lorazepam, alprazolam, etc.)
* herbal medications or preparations in doses designed to ameliorate nausea or emesis
* Patient has taken phenothiazines (prochlorperazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine, etc.) for any indication within the last 48 hours prior to the start of treatment with study drug
* Palonosetron is not permitted within 7 days prior to administration of investigational product
* Patient must not have been dosed with a test drug or blinded study drug in another investigational study within 30 days or 5 half-lives of the biologic activity of the test drug, whichever is longer, before the time of first study dose
* Patient who is receiving investigational agent(s) as part of another clinical study at the time of screening or who anticipates receiving investigational agent(s) during their scheduled radiotherapy and concomitant daily temozolomide therapy (Any exception to this criteria will be noted in a study Memo to File)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Affronti, DNP, RN, ANP, MHSc, Principal Investigator — The Preston Robert Tisch Brain Tumor Center at Duke
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 25 | 23
Completed | 22 | 21
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.56 (13.99) | 52.78 (13.95) | 52.67 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 21 | 45
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 22 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate as Measured by Antiemesis Tool (MAT)
Description: The Complete Response rate is defined as the proportion of participants with no emetic episode or the use of rescue medication during the first two weeks of radiation therapy and concomitant Temozolomide. The Complete Response rate will be assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT).
Time Frame: Weeks 1 and 2
Population: Four participants in each group did not complete MATs for the first two weeks.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
proportion of participants | 0.5717 | 0.7368
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Other; p = 0.2734, Chi-squared

2. Primary Outcome: Complete Response (CR) Rate as Measured by MAT With Supplemental Nurses Notes
Description: The Complete Response rate is defined as the proportion of participants with no emetic episode or the use of rescue medication during the first two weeks of radiation therapy and concomitant Temozolomide. The Complete Response rate will be assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) MAT and nurse notes if MATs are missing.
Time Frame: Weeks 1 and 2
Population: Forty participants completed MATs; data collected by nurses via telephone on the remaining 8 participants.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 25 | 23
proportion of participants | 0.6000 | 0.6522
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Other; p = 0.7091, Chi-squared

3. Secondary Outcome: Number of Participants Preferring Rolapitant in Combination With Ondansetron Versus Ondansetron Alone
Description: The number of participants who prefer rolapitant plus ondansetron over ondansetron alone, as determined by response to the question with "Which nausea medication regimen was I most satisfied with?"
Time Frame: Weeks 1-6
Population: Participants who provided treatment preference data.
Measure: Count of Participants; unit: Participants
Groups:
- Sequence A and Sequence B: Sequence A: Daily ondansetron alone for 3 weeks, followed by the use of rolapitant (one dose on day 22) plus continued daily ondansetron for 3 weeks.
  Sequence B: Single dose of rolapitant (one dose on day 1) plus daily ondansetron for 3 weeks, followed by daily ondansetron alone for 3 weeks.
  Rolapitant: single 180 mg dose by mouth
  Ondansetron: 8 mg by mouth daily
Arm/Group | Sequence A and Sequence B
Number analyzed (Participants) | 35
Participants
  Rolapitant + Ondansetron | 7
  Ondansetron alone | 21
  No Preference | 7
Statistical Analysis 1: Comparison: Sequence A and Sequence B; Test type: Equivalence — This was tested as patients who preferred rolapitant + ondansetron vs. patients who did not prefer rolapitant + ondansetron. Patients who reported no preference and preference to Ondansetron were combined; p = 0.0004, Exact Binomial
Statistical Analysis 2: Comparison: Sequence A and Sequence B; Test type: Equivalence — Three outcomes tested by sequence; p = 0.5207, Fisher Exact

4. Secondary Outcome: Week 3 Patient Satisfaction: Effectiveness
Description: Mean effectiveness scores at week 3 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The effectiveness subscale score was computed from the 3 items corresponding to effectiveness. The resulting effectiveness score is measured from 0-100 with higher scores corresponding to higher effectiveness.
Time Frame: Weeks 1-3
Population: Participants who responded to at least two of the TSQM-9 questions for the effectiveness subscale at week 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
score on a scale | 83.60 (20.14) | 94.44 (11.11)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Effectiveness during weeks 1-3 between sequences; p = 0.0406, t-test, 1 sided; T-test using the Satterthwaite method for unequal variances

5. Secondary Outcome: Week 3 Patient Satisfaction: Convenience
Description: Mean convenience scores at week 3 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The convenience subscale score was computed from the 3 items corresponding to convenience. The resulting convenience score is measured from 0-100 with higher scores corresponding to higher convenience.
Time Frame: Weeks 1-3
Population: Participants who responded to at least two of the TSQM-9 questions for the convenience subscale at week 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
score on a scale | 85.71 (15.57) | 94.15 (10.05)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Convenience during weeks 1-3 between sequences; p = 0.0541, t-test, 1 sided; T-test using the pooled method for equal variances

6. Secondary Outcome: Week 3 Patient Satisfaction: Overall Satisfaction
Description: Mean overall satisfaction scores at week 3 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The overall satisfaction subscale score was computed from the 3 items corresponding to overall satisfaction. The resulting overall satisfaction score is measured from 0-100 with higher scores corresponding to higher overall satisfaction.
Time Frame: Weeks 1-3
Population: Participants who responded to at least two of the TSQM-9 questions for the overall satisfaction subscale at week 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
score on a scale | 81.88 (17.69) | 90.94 (13.38)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Overall satisfaction during weeks 1-3 between sequences; p = 0.0781, t-test, 1 sided; T-test using the pooled method for equal variances

7. Secondary Outcome: Week 6 Patient Satisfaction: Effectiveness
Description: Mean effectiveness scores at week 6 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The effectiveness subscale score was computed by summing the 3 items corresponding to effectiveness. The resulting effectiveness score is measured from 0-100 with higher scores corresponding to higher effectiveness.
Time Frame: Weeks 4-6
Population: Participants who responded to at least two of the TSQM-9 questions for the effectiveness subscale at week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 20 | 18
score on a scale | 83.89 (17.28) | 88.27 (15.23)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Effectiveness during weeks 4-6 between sequences; p = 0.4146, t-test, 1 sided; T-test using the pooled method for equal variances

8. Secondary Outcome: Week 6 Patient Satisfaction: Convenience
Description: Mean convenience scores at week 6 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The convenience subscale score was computed from the 3 items corresponding to convenience. The resulting convenience score is measured from 0-100 with higher scores corresponding to higher convenience.
Time Frame: Weeks 4-6
Population: Participants who responded to at least two of the TSQM-9 questions for the convenience subscale at week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 20 | 18
score on a scale | 86.11 (16.07) | 91.98 (12.53)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Convenience during weeks 4-6 between sequences; p = 0.2214, t-test, 1 sided; T-test using the pooled method for equal variances

9. Secondary Outcome: Week 6 Patient Satisfaction: Overall Satisfaction
Description: Mean overall satisfaction scores at week 6 using the 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) patient satisfaction survey. The overall satisfaction subscale score was computed from the 3 items corresponding to overall satisfaction. The resulting overall satisfaction score is measured from 0-100 with higher scores corresponding to higher overall satisfaction.
Time Frame: Weeks 4-6
Population: Participants who responded to at least two of the TSQM-9 questions for the overall satisfaction subscale at week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 20 | 18
score on a scale | 81.39 (21.16) | 88.58 (12.12)
Statistical Analysis 1: Comparison: Sequence A vs Sequence B; Test type: Equivalence — Overall satisfaction during weeks 4-6 between sequences; p = 0.2028, t-test, 1 sided; T-test using the Satterthwaite method for unequal variances

10. Secondary Outcome: Chemoradiation-induced Nausea (cRIN) Rate Over First Two Weeks
Description: The cRIN-CR rate is defined as the proportion of participants who did not use rescue medication for nausea. The cRIN-CR rates were assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT).
Time Frame: Weeks 1 and 2
Population: Participants who completed MATs for the first two weeks.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
proportion of participants | 0.6160 | 0.6842

11. Secondary Outcome: Chemoradiation-induced Nausea (cRIN) Rate Over First Two Weeks and Supplemented by Nurses Notes
Description: The cRIN-CR rate is defined as the proportion of participants who did not use rescue medication for nausea. The cRIN-CR rates were assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT) and nurses notes if MATs were missing.
Time Frame: Weeks 1 and 2
Population: Forty participants completed MATs; data collected by nurses via telephone on the remaining 8 participants.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 25 | 23
proportion of participants | 0.6000 | 0.6087

12. Secondary Outcome: Chemoradiation-induced Vomiting (cRIV) Rate Over First Two Weeks
Description: The cRIV-CR rate is defined as the proportion of participants without use of rescue medication for vomiting. The cRIV-CR rates were assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT).
Time Frame: Weeks 1 and 2
Population: Participants who completed MATs for the first two weeks.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 21 | 19
proportion of participants | 0.8095 | 1.0000

13. Secondary Outcome: Chemoradiation-induced Vomiting (cRIV) Rate Over First Two Weeks With Supplemental Nurses Notes
Description: The cRIV-CR rate is defined as the proportion of participants without use of rescue medication for vomiting. The cRIV-CR rates were assessed via the modified Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT) and nurse notes if MATS are missing.
Time Frame: Weeks 1 and 2
Population: Forty participants completed MATs; data collected by nurses via telephone on the remaining 8 participants.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 25 | 23
proportion of participants | 0.8000 | 0.9565

14. Secondary Outcome: Chemoradiation-induced Nausea (cRIN) Rate Over All Six Weeks
Description: as for outcome 10
Time Frame: Weeks 1-6
Population: Participants who completed MATs for six weeks and complied with treatment.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 19 | 19
proportion of participants | 0.4737 | 0.4737

15. Secondary Outcome: Chemoradiation-induced Vomiting (cRIV) Rate Over All Six Weeks
Description: as for outcome 12
Time Frame: Weeks 1-6
Population: Data not collected on 10 participants.
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 19 | 19
proportion of participants | 0.7368 | 0.8947

16. Secondary Outcome: Ondansetron Medication Compliance Weeks 1-3
Description: Percentage of participants who adhered to ondansetron treatment for more than 21 days during weeks 1-3.
Time Frame: Weeks 1-3
Population: Participants who remained on study and returned medication logs.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 23 | 21
percentage of participants | 91.30 | 100

17. Secondary Outcome: Ondansetron Medication Compliance Weeks 4-6
Description: Percentage of participants who adhered to ondansetron treatment for more than 21 days during weeks 4-6.
Time Frame: Weeks 4-6
Population: Participants who remained on study without schedule changes and returned medication logs.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 20 | 21
percentage of participants | 95 | 95.24

18. Secondary Outcome: Proportion of Participants With Grade 3, 4 or 5 Treatment-related Adverse Events
Description: The proportion of participants with grade 3, 4 or 5 adverse events (severe, life-threatening, or fatal) possibly, probably or definitely related to administration of Rolapitant or Ondansetron. Adverse events will be collected from start of treatment through the end of the two-week period following chemoradiation (or until 30 days after the last dose of rolapitant is given in Sequence A). CTCAE version 4 was used to grade adverse events.
Time Frame: 8 weeks
Measure: Number; unit: proportion of participants
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 25 | 23
proportion of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Period 1 Rolapitant + Ondansetron: Weeks 1-3
  Rolapitant: single 180 mg dose by mouth
  Ondansetron: 8 mg by mouth daily
- Period 1 Ondansetron: Weeks 1-3
  Ondansetron: 8 mg by mouth daily
- Period 2 Rolapitant + Ondansetron: Weeks 4-6
  Rolapitant: single 180 mg dose by mouth
  Ondansetron: 8 mg by mouth daily
- Period 2 Ondansetron: Weeks 4-6
  Ondansetron: 8 mg by mouth daily
Arm/Group | Period 1 Rolapitant + Ondansetron | Period 1 Ondansetron | Period 2 Rolapitant + Ondansetron | Period 2 Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/23 | 0/25 | 1/22 | 2/23
Other Adverse Events (participants affected / at risk) | 22/23 | 23/25 | 18/22 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Rolapitant + Ondansetron (N=23) | Period 1 Ondansetron (N=25) | Period 2 Rolapitant + Ondansetron (N=22) | Period 2 Ondansetron (N=23)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 Rolapitant + Ondansetron (N=23) | Period 1 Ondansetron (N=25) | Period 2 Rolapitant + Ondansetron (N=22) | Period 2 Ondansetron (N=23)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 4 (4) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 6 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 9 (9) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Other, Specify: "muffling" in right ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other, Specify: ear fullness/muffling, hard to hear in both ears (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema Face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other, Specify: impaired vision, right eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other, Specify: right eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (8) | 12 (12) | 4 (4) | 3 (4)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other, Unspecified (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Other, Specify: constant feeling of being cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 4 (6) | 4 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Other, Specify: oral fungal infection on tongue (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 1 (7) | 1 (1) | 0 (0) | 1 (6)
Other, Specify: blurred vision preventing reading, d/t radiation mask placement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other, Specify: dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other, Specify: swollen eyelids impeding eye opening, d/t radiation mask placement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 3 (3) | 2 (3) | 9 (16) | 7 (10)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other, Specify: temporomandibular joint inflammation causing nausea while chewing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (11) | 11 (11) | 2 (2) | 7 (8)
Neck Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 2 (2) | 6 (11) | 5 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyramidal Tract Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Other, Specify: "bruising left hand from fall" (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
White Blood Cell Decreased (Investigations) | 2 (2) | 0 (0) | 3 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02991456/Prot_SAP_000.pdf